CLINICAL TRIAL: NCT01361893
Title: Factors Influencing the Racial Disparity in Sudden Infant Death Syndrome (SIDS)
Acronym: SIDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH); March of Dimes (Other)
Responsible Party: Principal Investigator, Rachel Moon, MD, Principal Investigator, Children's National Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 3488; K24RR023681 (NIH)
Record Dates: First submitted 2011-05-12; First posted 2011-05-27 (Estimated); Last update posted 2018-10-19 (Actual); Status verified 2018-10

CONDITIONS: Sudden Infant Death Syndrome
Keywords: SIDS; African American; Infants; Disparity
MeSH Terms: conditions — Sudden Infant Death | interventions — Evaluation Studies as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lifestyle Counseling (Other): Parents who qualify for the study will be asked to participate in the survey portion of the study. informed consent will be obtained. After completing the survey each parent will be asked if they would be willing to participate in and additional interview (focus group or semi-structured in-debth interview) at a later date.
  Interventions: Other: Lifestyle Counseling

INTERVENTIONS:
Other: Lifestyle Counseling — We will utilize a combination of quantitative and qualitative techniques to ascertain factors, attitudes, and beliefs of African American parents of infants less than 6 months old.
  Other Names: African American; Qualitative; Quantitative; SIDS; Infants

SUMMARY:
The overall purpose of this investigation is to better understand factors contributing to the high incidence of prone sleep positioning in African-American infants. In addition, the investigators are interested in investigating other races and ethinicities to understand their beliefs and perceptions and determine differences socioeconomically and socioculturally within and between groups. The investigators will address the following specific aims:

(-) To compare knowledge, attitudes, and practices regarding infant sleep position in parents of higher and lower SES.

(-) To identify risk factors for non-use of recommended supine sleep position in families with higher and lower SES (-) to develop a phenomenologic understanding of the decisions made by parents of higher SES and lower SES who do nt use recommended supine sleep position, using qualitative techniques.

DETAILED DESCRIPTION:
Epidemiologic studies have demonstrated prone position to be a major risk factor for SIDS. Studies have consistently demonstrated an increased rate of prone positioning in African American infants, but very little is known about the reasons why African American parents use the prone position more often than other racial groups. Furthermore, no studies have taken advantage of the observed socioeconomic status associated variablility in SIDS and prone sleeping within the African American community. By examing within-group differences, it is possible to move beyond comparative racial descriptions (i.e. comparisions of white and African American) to identification of potentially modifiable factors that might respond to culturally acceptable interventions within a disadvantaged group.

ELIGIBILITY:
Inclusion Criteria:

* Parents who are 18 years old wth children less than 6 months old are eligible to participate if they self-identify as African American, with parents born in the United States.

Exclusion Criteria:

* If the parent is male, not the custodial parent of the child, unable to complet the interview in English or if their child has a chronis illness that would preclude use of the supine sleep position, severe gastroesophageal reflux or recent spinal surgery.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 616 (Actual)
Dates: Start 2004-12; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Factors Influencing the Racial Disparity in SIDS | December 2004 - June 2011
  Sleep Position (Supine vs. Nonsupine) Bedsharing (Yes vs. No) Use of Softbedding (Yes vs. No)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Y Moon, MD, Principal Investigator — University of Virginia
Locations (1):
- Children's National Medical Center, Washington D.C., District of Columbia, United States